CLINICAL TRIAL: NCT02493374
Title: Mitigation of Type 2 Diabetes in Hypercholesterolemic Patients Undergoing a Partial Ileal Bypass
Brief Title: Mitigation of Type 2 Diabetes by Partial Ileal Bypass
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: University of Minnesota (Other)
Collaborators: Weill Medical College of Cornell University (Other); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1504M69662
Record Dates: First submitted 2015-07-06; First posted 2015-07-09 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a study of people with type 2 diabetes and high cholesterol between age 18 and 65. This study is trying to figure out if a partial bypass of the small intestine can reverse type 2 diabetes for people who require cholesterol lowering and who cannot tolerate the statin drugs.

DETAILED DESCRIPTION:
The partial ileal bypass (PIB) operation is a standard procedure used in the management of hyperlipidmia since 1963. POSCH was the intervention modality in the National Institutes of Health, National Heart Lung and Blood Institute-funded Program on the Surgical Control of the Hyperlipidemias (POSCH) trial. The POSCH study was a secondary trial in patients with a documented prior myocardial infarction. The trial compared the post-dietary lipid therapy changes in 421 PIB-intervention patients to 417 controls, with a lowering of total plasma cholesterol of 24% (P<0.0001), a lowering of low density lipoprotein (LDL)-cholesterol of 38% (P<0.0001), and an elevation of high density lipoprotein (HDL)-cholesterol of 4% (P=0.02). These lipid changes were associated with a 35% (P<0.001) reduction in the intervention group of death due to coronary heart disease and confirmed recurrent myocardial infarction, as well as a 27% (P<0.038) reduction in peripheral vascular disease, and a 54% (P<0.005) diminution in the occurrence of coronary artery surgery or angioplasty. Concurrently with the clinical study, POSCH assessed sequential coronary arteriograms at 0, 3, 5, 7, and 10 years, which showed less disease progression in the surgery group, and even statistically significant plaque regression in the PIB cohort. POSCH PIB patients exhibited a statistically significant increase in life expectancy; this finding persisted at a 25-year follow-up assessment.

In the field of metabolic/bariatric surgery, resolution of type 2 diabetes by gastrointestinal tract manipulations was clearly demonstrated by 1998. In three meta-analyses, the procedures that involved shortening of the ileum (biliopancreatic diversion and duodenal switch) were responsible for the highest percentage of type 2 diabetes resolution. Recently under evaluation are standard metabolic/bariatric and experimental metabolic operations that will engender type 2 diabetes resolution with minimal or no weight loss in non-obese diabetic patients.

The gut-diabetes relationship has often been attributed to an increased elaboration of the hormones glucagon-like peptide-1 (GLP-1) and peptide YY (PYY), both secreted by the L-cells of the intestinal mucosa. These hormones seem to work in concert, either eliciting the same metabolic response or augmenting the actions of the other. With respect to pancreatic endocrine function, GLP-1 and PYY contribute to the incretin effect, counteract the insulin depression action of gastrin stimulating peptide and gastrin-releasing peptide, and stimulate glucose-dependent insulin secretion, preinsulin gene expression, beta-cell proliferation, and antiapoptopic pathways. It has been shown that GLP-1 secretion is reduced in patients with type 2 diabetes. In a recent study of the effects of direct human terminal ileum and cecal contact with a food hydrolysate, significant plasma GLP-1 and PYY elevations were demonstrated, confirming the ability of the cecum, as well as the ileum, to secrete GLP-1 and PYY on stimulation. In the Goto-Kakizaki rat with naturally occurring type 2 diabetes, ileal bypass or excision did not lower GLP-1 production, but interestingly increased it five- to six-fold.

These complementary studies gave rise to the hypothesis that: the PIB operation, in addition to its action on cholesterol metabolism, may aslo prevent and resolve type 2 diabetes.

In our laboratory at the University of Minnesota, the investigators have clearly established the mechanism for the reduction of total cholesterol and LDL-cholesterol by PIB: interference with the cholesterol and bile acid enterohepatic cycles, markedly decreased absorption and reabsorption of cholesterol and bile acids, increased excretion of cholesterol and bile acids, increased turnover of cholesterol to generate bile acids and replenish the cholesterol pool, and the insufficient ability of the body (even in familial hypercholesterolemics) to maintain the miscible (plasma and liver) and less-freely miscible (tissues, including the arteries) body pools, and, thereby, a depletion of the cholesterol content of atherosclerotic plaques. the investigators have now (see above) added to that knowledge that the elimination of the terminal ileum from the intestinal pathway will increase circulating GLP-1 levels, with this incretin probably emanating from the cecum.

The investigators have now completed and submitted for publication our study on the incidence of type 2 diabetes in the POSCH program 25 plus years after formal trial closure (IRB Code Number: 1408M53283). The title of our paper is "Partial Ileal Bypass Affords Protection from Onset of Type 2 Diabetes". Of the 66 control patient responders in POSCH, 17 contracted type 2 diabetes (25.8%); of 80 PIB responders, 8 contracted type 2 diabetes (10%). The difference between groups was significant (P=0.015 by Fisher Exact Test) with an odds ratio of 0.320 for the PIB group and an over two-fold (2.6) increase in the incidence of type 2 diabetes in the controls. Including borderline type 2 diabetes (prediabetic) patients, these values were 22 of 66 controls (33.3%) and 10 of 80 PIB patients (12.5%), with an odds ratio of 0.286 and a P<0.004, and again an over two-fold (2.7) increase in the incidence of type 2 diabetes in the control patients. Therefore, PIB appeared to afford protection from the onset of type 2 diabetes for over 30 years.

ELIGIBILITY:
Inclusion Criteria:

* Hyperlipidemia patients referred for partial ileal bypass, who also have type 2 diabetes.

Exclusion Criteria:

* Preoperative C-peptide indicative of non-functioning islet cells.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals in need of lipid modification but are intolerant of statin drugs who are referred for a partial ileal bypass (PIB) operation, still the most efficacious means to treat hyperlipidemia. In the subgroup of these patients who also have type 2 diabetes, with a functioning pancreas, we hope to perform a pilot study on the effect of PIB on type 2 diabetes.
  Study blood tests:
  - Pre-PIB and at 6 month and 12 months postop fasting blood samples for glucose, hemoglobin A1c, insulin, C-peptide, GLP-1, ghrelin, and glucagon; then after oral glucose meal testing for determination of glucose, GLP-1, and ghrelin at 30, 60, 90, and 120 minutes.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Mitigation of Type 2 Diabetes | 3 years
  Blood draws only

CONTACTS AND LOCATIONS:
Overall Officials: Henry Buchwald, MD, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided